CLINICAL TRIAL: NCT06742463
Title: Venetoclax Combined With HAG Regimen in Treating Adult Relapse/Refractory Acute T Cell Lymphoblastic Leukemia/Lymphoma: A Phase II, Single Arm and Multicenter Study
Brief Title: VHAG in Treating R/R T-ALL/LBL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20240113C
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-10

CONDITIONS: Acute T Lymphpblastic Leukemia/Lymphoma
Keywords: acute lymphoblastic leukemia; chemotherapy; relapse; refractory
MeSH Terms: conditions — Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence | interventions — venetoclax; Homoharringtonine; Cytarabine; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Venetoclax for 4weeks(adjust according to BM on Day15), oral; Homoharringtonine for 1 week,iv; Cytarabine for 10-14 dsys, sc; G-CSF.
  Interventions: Drug: Venetoclax; Drug: homoharringtonine; Drug: Cytarabine (Ara-C); Drug: G-CSF

INTERVENTIONS:
Drug: Venetoclax — BCL-2 inhibitor
Drug: homoharringtonine — alkaloid
Drug: Cytarabine (Ara-C) — Metabolic antagonist.
Drug: G-CSF — Granulocyte colony-stimulating factor

SUMMARY:
Acute T cell lymphoblastic leukemia/lymphoma (T-ALL/LBL) is an aggressive type of leukemia that results from the malignant evolution of T-lineage progenitor cells at different differentiation stages. After induction chemotherapy and consolidation chemotherapy, there are still about 30% of patients who cannot achieve complete remission of clinical symptoms or negative MRD. This is also an important factor for the recurrence of ALL patients. In addition, most relapsed T-ALL/LBL patients relapse during first-line treatment. Once the disease relapses, it is difficult to cure for most young and adult patients, and the overall survival rate of patients is less than 10%.

DETAILED DESCRIPTION:
This is a prospective, single-arm, phase II and open-label study. A total of 50 R/R T-ALL/LBL participants will be enrolled. The primary endpoint is complete remission with or without peripheral blood cell recovery. The induction therapy is a combination of Venetoclax(Ven), Homoharringtonine(HHT) , Cytarabine and G-CSF. The purpose of this study is to explore efficacy of the VHAG in the treatment of R/R T-ALL/LBL patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Before enrollment, a diagnosis of newly diagnosed T-cell acute leukemia/lymphoma.The diagnostic criteria refer to the 2022 WHO classification; 2. Age ≥ 14 years,<75 years; 3. Clincally diagnosed as relapsed or refractory T-ALL/LBL; 4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2; 5. Expected survival time ≥ 2 months; 6. No organ dysfunction that would restrict the use of this protocol during the screening period; 7. Understand the study and sign the informed consent form.

Exclusion Criteria:

* 1. Patients with known central nervous system (CNS) involvement of T-ALL/LBL; 2. Diseases with abnormal heart, lung, liver, kidney, or other organ functions that may limit the patient's participation in this trial (including but not limited to severe infections, uncontrolled diabetes, severe heart failure or angina, active pulmonary tuberculosis, asthma, COPD, bronchiectasis, etc.) 3. Cardiac ultrasound LVEF < 45%; 4. History of other malignancies within the past 5 years, excluding localized thyroid cancer and in situ skin cancer; 5. Serum total bilirubin > 1.5 ULN (upper limit of normal); ALT or AST > 2.5 ULN; serum creatinine > 1.5 ULN; 6. Known HIV infection; 7. Conditions affecting the use of the study drug as assessed by the investigator; 8. Inability to understand or comply with the study protocol.

Ages: 14 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Complete remission with or without incomplete PB cell recovery(CR/CRi) rate | at the end of Cycle 1 and 2（each cycle is 28days）
  Blast rate lower than 5% with or without peripheral blood cell recovery

SECONDARY OUTCOMES:
Overall survival (OS) | up to 5 years
  Defined for all patients in a trial; measured from day 1 of treatment to the date of death from any cause;
Event free survival(EFS) | up to 2 years
  Defined for all patients in a trial; measured from day 1 of treatment to the date of treatment failure, hematologic relapse from CR/CRi or death from any cause, whichever occurs first;
Minimal residual disease (MRD) | At the end of Cycle 1 and 2（each cycle is 28 days）
  MRD level detected by flow cytometry which value <0.1% is defined as negtive
Adverse event | At the end of Cycle 1 and 2
  Safety of induction therapy

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peirs S, Matthijssens F, Goossens S, Van de Walle I, Ruggero K, de Bock CE, Degryse S, Cante-Barrett K, Briot D, Clappier E, Lammens T, De Moerloose B, Benoit Y, Poppe B, Meijerink JP, Cools J, Soulier J, Rabbitts TH, Taghon T, Speleman F, Van Vlierberghe P. ABT-199 mediated inhibition of BCL-2 as a novel therapeutic strategy in T-cell acute lymphoblastic leukemia. Blood. 2014 Dec 11;124(25):3738-47. doi: 10.1182/blood-2014-05-574566. Epub 2014 Oct 9. PMID 25301704
- [Background] Stock W, Luger SM, Advani AS, Yin J, Harvey RC, Mullighan CG, Willman CL, Fulton N, Laumann KM, Malnassy G, Paietta E, Parker E, Geyer S, Mrozek K, Bloomfield CD, Sanford B, Marcucci G, Liedtke M, Claxton DF, Foster MC, Bogart JA, Grecula JC, Appelbaum FR, Erba H, Litzow MR, Tallman MS, Stone RM, Larson RA. A pediatric regimen for older adolescents and young adults with acute lymphoblastic leukemia: results of CALGB 10403. Blood. 2019 Apr 4;133(14):1548-1559. doi: 10.1182/blood-2018-10-881961. Epub 2019 Jan 18. PMID 30658992
- [Background] Dunsmore KP, Winter SS, Devidas M, Wood BL, Esiashvili N, Chen Z, Eisenberg N, Briegel N, Hayashi RJ, Gastier-Foster JM, Carroll AJ, Heerema NA, Asselin BL, Rabin KR, Zweidler-Mckay PA, Raetz EA, Loh ML, Schultz KR, Winick NJ, Carroll WL, Hunger SP. Children's Oncology Group AALL0434: A Phase III Randomized Clinical Trial Testing Nelarabine in Newly Diagnosed T-Cell Acute Lymphoblastic Leukemia. J Clin Oncol. 2020 Oct 1;38(28):3282-3293. doi: 10.1200/JCO.20.00256. Epub 2020 Aug 19. PMID 32813610
- [Background] Quist-Paulsen P, Toft N, Heyman M, Abrahamsson J, Griskevicius L, Hallbook H, Jonsson OG, Palk K, Vaitkeviciene G, Vettenranta K, Asberg A, Frandsen TL, Opdahl S, Marquart HV, Siitonen S, Osnes LT, Hultdin M, Overgaard UM, Wartiovaara-Kautto U, Schmiegelow K. T-cell acute lymphoblastic leukemia in patients 1-45 years treated with the pediatric NOPHO ALL2008 protocol. Leukemia. 2020 Feb;34(2):347-357. doi: 10.1038/s41375-019-0598-2. Epub 2019 Oct 14. PMID 31611626
- [Background] Chiaretti S, Vitale A, Cazzaniga G, Orlando SM, Silvestri D, Fazi P, Valsecchi MG, Elia L, Testi AM, Mancini F, Conter V, te Kronnie G, Ferrara F, Di Raimondo F, Tedeschi A, Fioritoni G, Fabbiano F, Meloni G, Specchia G, Pizzolo G, Mandelli F, Guarini A, Basso G, Biondi A, Foa R. Clinico-biological features of 5202 patients with acute lymphoblastic leukemia enrolled in the Italian AIEOP and GIMEMA protocols and stratified in age cohorts. Haematologica. 2013 Nov;98(11):1702-10. doi: 10.3324/haematol.2012.080432. Epub 2013 May 28. PMID 23716539